CLINICAL TRIAL: NCT00017394
Title: A Phase II Study of Bevacizumab in Combination With Vinorelbine in Stage IV Breast Cancer
Brief Title: Bevacizumab Plus Vinorelbine in Treating Patients With Stage IV Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02388; 01-013; CDR0000068685 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-06-06; First posted 2003-06-12 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Male Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — Bevacizumab; Vinorelbine

ARMS (1):
- Treatment (bevacizumab, vinorelbine tartrate) (Experimental): Patients receive bevacizumab IV over 30-90 minutes once every other week and vinorelbine IV over 6-10 minutes once weekly for 8 weeks. Treatment repeats every 8 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Patients with complete or partial response or stable disease after completion of the fourth course may receive additional courses of concurrent bevacizumab and vinorelbine administered once every other week or may continue therapy on the schedule as above.
  Interventions: Biological: bevacizumab; Drug: vinorelbine tartrate; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Drug: vinorelbine tartrate — Given IV
  Other Names: Eunades; navelbine ditartrate; NVB; VNB
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of bevacizumab combined with vinorelbine in treating patients who have stage IV breast cancer. Monoclonal antibodies such as bevacizumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining monoclonal antibody with chemotherapy may kill more cancer cells

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the complete and partial response rates in patients with stage IV breast cancer treated with concurrent bevacizumab and vinorelbine.

II. Determine the side effects of this regimen in these patients. III. Determine the time to disease progression in patients treated with this regimen.

IV. Determine the time on study (a reflection of time to progression, treatment-related side effects, and patient preference) of patients treated with this regimen.

V. Assess urine protein/creatinine ratio and serum complement levels as screening measures for renal injury in patients treated with bevacizumab.

OUTLINE: This is a multicenter study.

Patients receive bevacizumab IV over 30-90 minutes once every other week and vinorelbine IV over 6-10 minutes once weekly for 8 weeks. Treatment repeats every 8 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Patients with complete or partial response or stable disease after completion of the fourth course may receive additional courses of concurrent bevacizumab and vinorelbine administered once every other week or may continue therapy on the schedule as above.

PROJECTED ACCRUAL: A total of 56 patients will be accrued for this study within 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed stage IV breast cancer

  * Patients without pathologic or cytologic confirmation of metastatic disease must have unequivocal evidence of metastasis by physical exam or radiologic study
* Must meet 1 of the following criteria:

  * Received 1 or 2 prior conventional chemotherapy regimens for metastatic disease
  * Relapsed within 1 year after adjuvant chemotherapy and no prior chemotherapy for metastatic disease
* At least 1 unidimensionally measurable lesion, meeting 1 of the following criteria:

  * At least 20 mm by conventional techniques
  * At least 10 mm by spiral CT scan
* No CNS metastases by CT scan or MRI within the past 6 weeks
* No prior or concurrent primary CNS tumor on physical exam
* Disease progression after bone marrow or peripheral blood stem cell transplantation allowed
* HER2-positive tumors allowed if previously treated with trastuzumab (Herceptin)
* Hormone receptor status:

  * Not specified
* Male or female
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* More than 3 months
* Absolute neutrophil count at least 1,500/mm^3
* Hemoglobin at least 9 g/dL
* Platelet count at least 100,000/mm^3
* No prior bleeding diathesis or coagulopathy
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST/ALT no greater than 2.5 times ULN
* INR no greater than 1.5
* Creatinine less than 2 mg/dL
* Urine protein no greater than +1 by dipstick
* Urine protein less than 500 mg by 24-hour urine collection
* LVEF at least 50%
* No prior stroke
* No New York Heart Association class II-IV congestive heart failure
* No serious cardiac arrhythmia requiring medication, including atrial fibrillation requiring systemic anticoagulation
* No grade II or greater peripheral vascular disease within the past year
* No clinically significant peripheral artery disease
* No deep vein thrombosis or embolism within the past 5 years
* No arterial thromboembolic event within the past 6 months, including any of the following:

  * Transient ischemic attack
  * Cerebrovascular accident
  * Unstable angina
  * Myocardial infarction
* No other significant cardiovascular disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No evidence of seizures not controlled with standard medical therapy
* No prior allergic reactions attributed to compounds of similar chemical or biologic composition to bevacizumab or other agents used in the study
* Prior mild infusion reaction to trastuzumab allowed
* No serious non-healing wound, ulcer, or bone fracture
* No significant traumatic injury within the past 4 weeks
* No other concurrent illness (such as active infection) that would require active treatment or preclude study
* No psychiatric illness or social situation that would preclude study
* See Disease Characteristics
* No prior bevacizumab
* No other prior experimental angiogenesis inhibitors
* At least 2 weeks since prior trastuzumab and recovered
* Concurrent epoetin alfa or filgrastim (G-CSF) allowed
* See Disease Characteristics
* At least 2 weeks since prior chemotherapy and recovered
* No prior vinorelbine
* No more than 2 prior conventional chemotherapy regimens for metastatic breast cancer
* Prior hormonal therapy allowed
* At least 1 week since prior radiotherapy and recovered
* No concurrent radiotherapy
* At least 4 weeks since prior major surgical procedure or open biopsy
* At least 1 week since prior fine-needle aspiration except in the breast
* No concurrent major surgical procedure
* Recovered from the toxic effects of any prior therapy
* At least 10 days since prior oral or parenteral anticoagulants (e.g., heparin or warfarin) except to maintain the patency of permanent, indwelling central venous catheter
* At least 10 days since prior thrombolytic agents
* No chronic aspirin therapy greater than 325 mg per day or non-steroidal anti-inflammatory medications that inhibit platelet function
* No concurrent COX-2 inhibitors that inhibit platelet function
* No other concurrent investigational or commercial agents or therapies for the malignancy
* No concurrent antiretroviral therapy for HIV-positive patients
* No concurrent ketoconazole, zidovudine, or macrolide antibiotics
* No concurrent oral or parenteral anticoagulants except to maintain patency of permanent, indwelling central venous catheter
* No concurrent thrombolytic agent
* Concurrent bisphosphonates allowed
* Concurrent celecoxib or rofecoxib allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2001-03; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Response rate to combination therapy with bevacizumab and vinorelbine, defined by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria | Up to 6 years

SECONDARY OUTCOMES:
Time to progression | Time from the first treatment on study until the time of documented disease progression, assessed up to 6 years
Toxicities, graded according to the National Cancer Institute Common Toxicity Criteria (NCI CTC) v2.0 | Up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Harold Burstein, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States